CLINICAL TRIAL: NCT02737826
Title: Discontinuation From Chronic Opioid Therapy For Pain Using a Buprenorphine Taper
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Pro00046473
Record Dates: First submitted 2016-03-14; First posted 2016-04-14 (Estimated); Results first posted 2021-04-13 (Actual); Last update posted 2022-12-01 (Actual); Status verified 2022-11

CONDITIONS: Chronic Pain; Opioid Pain Medication
MeSH Terms: conditions — Chronic Pain | interventions — Gabapentin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Phase - Buprenorphine Initiation (Experimental): In Phase I, we will determine buprenorphine tolerability using a one-day outpatient buprenorphine initiation protocol up to 16mg sublingually over an up to 8 hour induction window. "Buprenorphine tolerability" will be defined as pain level ≤ to baseline, withdrawal measures ≤ to baseline, and willingness to continue with taper.
  Interventions: Drug: Buprenorphine Initiation - Phase I
- Phase II - Gabapentin + Buprenorphine (Active Comparator): Subjects who tolerate sublingual buprenorphine initiation in Phase I will proceed to Phase II, which will involve randomization to gabapentin or placebo, 2 week stabilization period, and up to 8 week buprenorphine tapering period. Those randomized to gabapentin will receive up to 1600mg oral gabapentin (double blinded) divided three times daily, titrated over the 2 week stabilization period and continued during the buprenorphine tapering period. During the 2 week stabilization period, buprenorphine will also be titrated up to 24mg as needed/tolerated.
  Interventions: Drug: Gabapentin + Buprenorphine - Phase II
- Phase II - Placebo + Buprenorphine (Placebo Comparator): Subjects who tolerate sublingual buprenorphine initiation in Phase I will proceed to Phase II, which will involve randomization to gabapentin or placebo, 2 week stabilization period, and up to 8 week buprenorphine tapering period. Those randomized to placebo will receive up to 1600mg oral placebo (double blinded) divided three times daily, titrated over the 2 week stabilization period and continued during the buprenorphine tapering period. During the 2 week stabilization period, buprenorphine will also be titrated up to 24mg as needed/tolerated.
  Interventions: Drug: Placebo + Buprenorphine - Phase II
- Phase II - Buprenorphine taper (Experimental): After a 2 week stabilization period where sublingual buprenorphine is titrated up to 24 mg/day and oral gabapentin/placebo is titrated up to 1600mg/day, subjects will enter a buprenorphine tapering period lasting up to 8 weeks. The suggested buprenorphine taper will be determined by stabilizing dose, but able to be altered by prescriber or participant based on symptoms.
  Interventions: Drug: Buprenorphine taper - Phase II

INTERVENTIONS:
Drug: Buprenorphine Initiation - Phase I — In Phase I, we will determine buprenorphine tolerability using a one-day outpatient buprenorphine initiation protocol up to 16mg sublingually over an 8 hour induction window.
  Arms: Phase - Buprenorphine Initiation
Drug: Gabapentin + Buprenorphine - Phase II — Subjects who tolerate sublingual buprenorphine initiation in Phase I will proceed to Phase II, which will involve randomization to oral gabapentin or placebo, 2 week stabilization period, and up to 8 week buprenorphine tapering period. Those randomized to gabapentin will receive up to 1600mg gabapentin (double blinded) divided three times daily, titrated over the 2 week stabilization period and continued during the buprenorphine tapering period. During the 2 week stabilization period, buprenorphine will also be titrated up to 24mg as needed/tolerated.
  Arms: Phase II - Gabapentin + Buprenorphine
Drug: Placebo + Buprenorphine - Phase II — Subjects who tolerate sublingual buprenorphine initiation in Phase I will proceed to Phase II, which will involve randomization to oral gabapentin or placebo, 2 week stabilization period, and up to 8 week buprenorphine tapering period. Those randomized to placebo will receive up to 1600mg placebo (double blinded) divided three times daily, titrated over the 2 week stabilization period and continued during the buprenorphine tapering period. During the 2 week stabilization period, buprenorphine will also be titrated up to 24mg as needed/tolerated.
  Arms: Phase II - Placebo + Buprenorphine
Drug: Buprenorphine taper - Phase II — After a 2 week stabilization period where sublingual buprenorphine is titrated up to 24 mg/day and oral gabapentin/placebo is titrated up to 1600mg/day, subjects will enter a buprenorphine tapering period lasting up to 8 weeks. The suggested buprenorphine taper will be determined by stabilizing dose, but able to be altered by prescriber or participant based on symptoms.
  Arms: Phase II - Buprenorphine taper

SUMMARY:
Chronic opioid therapy for pain can be associated with significant risks, and a significant number of patients maintained on chronic opioids have continued pain and/or poor functioning. When patients need to or want to come off their opioid pain medications, there is little to guide physicians as to how to best help them do so, and it is not known how patients do after coming off opioid medications. The goals of this study are (1) to evaluate two medications in assisting patients in coming off their opioid pain medications and (2) determining outcomes after discontinuing opioids.

ELIGIBILITY:
Inclusion Criteria:

* 18 - 70 years of age
* Ability to speak and read in English
* Currently taking chronic opioid therapy for pain for at least 6 months
* On opioid dose of >60mg and <200mg oral morphine equivalents/day
* Voluntarily seeking opioid discontinuation
* Willing to attempt buprenorphine-assisted opioid discontinuation
* Willing to be randomized to gabapentin or placebo
* Have current physician who is actively prescribing opioids and who will be notified by the research team of the patient's entry into the study.

Exclusion Criteria:

* Previous intolerance or allergy to buprenorphine or gabapentin
* Diagnostic & Statistical Manual -V criteria for substance use disorder currently or in the past (other than nicotine)
* Unstable medical or psychiatric condition that would preclude safe or meaningful participation (e.g. traumatic brain injury; severe mental illness; severe cardiac, renal, pulmonary, or liver disease)
* Current use of illicit drugs
* Maintenance on fentanyl or methadone
* Current treatment with gabapentin

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2019-12-09 (Actual); Study Completion 2021-01-13 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase I - Buprenorphine Initiation: In Phase I, we will determine buprenorphine tolerability using a one-day outpatient buprenorphine initiation protocol using up to 16mg of buprenoprhine over an up to 8 hour induction window. "Buprenorphine tolerability" will be defined as pain level ≤ to baseline, withdrawal measures ≤ to baseline, and willingness to continue with taper.
  Buprenorphine - Phase I: In Phase I, we will determine buprenorphine tolerability using a one-day outpatient buprenorphine initiation protocol.
- Phase II - Gabapentin + Buprenorphine Taper: Subjects who tolerate buprenorphine initiation in Phase I (determined by pain level ≤ to baseline, withdrawal measures ≤ to baseline, and willingness to continue with taper) will proceed to Phase II, which will involve randomization to gabapentin or placebo, 2 week stabilization period where buprenorphine will be titrated up as tolerated/needed to a maximum of 24 mg/day and gabapentin will be titrated up to 1600mg/day in 3 daily doses as tolerated. After the 2 week stabilization period, buprenorphine tapering will begin according to a tapering schedule that will last up to 8 weeks based on stabilizing buprenorphine dose.
  After the buprenorphine taper is complete, a 1 week taper of gabapentin will be provided.
- Phase II - Placebo + Buprenorphine Taper: Subjects who tolerate buprenorphine initiation in Phase I (determined by pain level ≤ to baseline, withdrawal measures ≤ to baseline, and willingness to continue with taper) will proceed to Phase II, which will involve randomization to gabapentin or placebo, 2 week stabilization period where buprenorphine will be titrated up as tolerated/needed to a maximum of 24 mg/day and placebo will be titrated up to 1600mg/day in 3 daily doses as tolerated. After the 2 week stabilization period, buprenorphine tapering will begin according to a tapering schedule that will last up to 8 weeks based on stabilizing buprenorphine dose.
  After the buprenorphine taper is complete, a 1 week taper of placebo will be provided.
Period: Phase I - Buprenorphine Initiation
Arm/Group | Phase I - Buprenorphine Initiation | Phase II - Gabapentin + Buprenorphine Taper | Phase II - Placebo + Buprenorphine Taper
Started | 27 | 0 | 0
Completed | 27 | 0 | 0
Not Completed | 0 | 0 | 0
Period: Phase II - Randomization + Taper
Arm/Group | Phase I - Buprenorphine Initiation | Phase II - Gabapentin + Buprenorphine Taper | Phase II - Placebo + Buprenorphine Taper
Started | 0 | 13 | 14
Completed | 0 | 1 | 0
Not Completed | 0 | 12 | 14
Not completed — Withdrawal by Subject | 0 | 12 | 14

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: In Phase I, we will determine buprenorphine tolerability using a one-day outpatient buprenorphine initiation protocol. "Buprenorphine tolerability" will be defined as pain level ≤ to baseline, withdrawal measures ≤ to baseline, and willingness to continue with taper.
  Buprenorphine - Phase I: In Phase I, we will determine buprenorphine tolerability using a one-day outpatient buprenorphine initiation protocol.
Arm/Group | All Study Participants
Number analyzed (Participants) | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.48 (11.11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 26
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 19
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 27

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients Who Tolerate Buprenorphine Initiation
Description: For Phase I, the primary outcome measure is the percentage of patients who tolerate buprenorphine initiation within an 8-hour initiation period, as evidenced by a total score of 3 points when summing the following measures (1) moderate-good level of pain control (same or improved rating on a 0-10 visual analogue scale for pain) = 1 point, (2) mild to no withdrawal symptoms (≤10 on the Subjective Opioid Withdrawal Scale) = 1 point, and (3) willingness to continue to the stabilization and tapering phase of the study; "yes" = 1 point.
Time Frame: 8 hours post dose
Measure: Count of Participants; unit: Participants
Groups:
- Phase I - Buprenorphine Initiation: In Phase I, we will determine buprenorphine tolerability using a one-day outpatient buprenorphine initiation protocol. "Buprenorphine tolerability" will be defined as pain level ≤ to baseline, withdrawal measures ≤ to baseline, and willingness to continue with taper.
  Buprenorphine - Phase I: In Phase I, we will determine buprenorphine tolerability using a one-day outpatient buprenorphine initiation protocol.
Arm/Group | Phase I - Buprenorphine Initiation
Number analyzed (Participants) | 27
Participants | 27

2. Primary Outcome: Number of Participants Who Achieve Opioid Cessation
Description: For Phase II, the primary outcome measure will be number of participants opioid who achieve cessation 8 weeks after stabilization at Week 10, evidenced as a score of 3 points when summing the following measures: self-report of no opioid use = 1 point; prescription drug monitoring data showing no opioid prescriptions filled in past 30 days = 1 point; and confirmatory negative urine toxicology for a full panel of opioids = 1 point.
Time Frame: 8 weeks after stabilization at Week 10
Measure: Count of Participants; unit: Participants
Groups:
- Phase II - Gabapentin + Buprenorphine Taper; Phase II - Placebo + Buprenorphine Taper: Subjects who tolerate buprenorphine initiation in Phase I (determined by pain level ≤ to baseline, withdrawal measures ≤ to baseline, and willingness to continue with taper) will proceed to Phase II, which will involve randomization to gabapentin or placebo, buprenorphine stabilization, and buprenorphine tapering.
  Buprenorphine - Phase I: In Phase I, we will determine buprenorphine tolerability using a one-day outpatient buprenorphine initiation protocol.
  Gabapentin - Phase II: Subjects who tolerate buprenorphine initiation (determined by pain level ≤ to baseline, withdrawal measures ≤ to baseline, and willingness to continue with taper) will proceed to Phase II, which will involve randomization to gabapentin or placebo, buprenorphine stabilization, and buprenorphine tapering.
  Placebo - Phase II: Subjects who tolerate buprenorphine initiation (determined by pain level ≤ to baseline, withdrawal measures ≤ to baseline, and willingness to continue with taper) will proceed to Phase II, which will involve randomization to gabapentin or placebo, buprenorphine stabilization, and buprenorphine tapering.
Arm/Group | Phase II - Gabapentin + Buprenorphine Taper | Phase II - Placebo + Buprenorphine Taper
Number analyzed (Participants) | 13 | 14
Participants | 1 | 0

3. Secondary Outcome: Number of Participants Who Achieve Opioid Cessation Post-taper: 1 Month
Description: Opioid cessation post taper: 1 month with opioid cessation measured through self-report, prescription drug monitoring data, and confirmatory UDS for a full panel of opioids.
Time Frame: 1 month post-taper
Population: Only one person in the Gabapentin + Buprenorphine Taper Arm completed the 8 week study buprenorphine taper, making them eligible for analysis for this secondary outcome measure. Zero people in the Placebo + Buprenorphne Taper Arm completed the study buprenorphine taper.
Measure: Count of Participants; unit: Participants
Groups:
- Gabapentin + Buprenorphine Taper - Opioid Cessation 1 Month Post-taper: One person in the Gabapentin + Buprenorphine Taper Arm completed the study buprenorphine taper
- Placebo + Buprenorphine Taper - Opioid Cessation 1 Month Post-taper: Zero persons in the Placebo + Buprenorphine Taper Arm completed the study buprenorphine taper.
Arm/Group | Gabapentin + Buprenorphine Taper - Opioid Cessation 1 Month Post-taper | Placebo + Buprenorphine Taper - Opioid Cessation 1 Month Post-taper
Number analyzed (Participants) | 1 | 0
Participants | 0 | 0

4. Secondary Outcome: Pain Self-report: Pain Catastrophizing Scale - Baseline
Description: The Self Reporting Pain Catastrophizing scale consists of 13 items scored from 0 to 4. The total possible score is 52. A higher score indicates more catastrophizing thoughts are present. A lower score indicates less catastrophizing thoughts.
Time Frame: Baseline
Population: One consented and randomized participant in the Placebo + Buprenorphine Taper Arm was erroneously randomized prior to buprenorphine induction, and dropped out of the study on the day of induction prior to receiving first buprenorphine dose (prior to eligibility for randomization). This participant is not included in this analysis.
Measure: Mean (Full Range); unit: units on a scale
Groups:
- Gabapentin + Buprenorphine Taper; Placebo + Buprenorphine Taper: N=13 in this arm
Arm/Group | Gabapentin + Buprenorphine Taper | Placebo + Buprenorphine Taper
Number analyzed (Participants) | 13 | 13
units on a scale | 21.9 [3 to 39] | 21.2 [0 to 48]

5. Secondary Outcome: Pain Laboratory Testing: Mechanical - Baseline
Description: Mechanical (Pressure) Pain Threshold Assessment (PPTh): A digital anesthesiometer (IITC Life Sciences ElectroVonFrey) will be used to assess mechanical pain perception. Pain threshold to static mechanical stimuli will be determined by applying the rigid monofilament to the dorsum of each subject's right hand with increasing pressure (10 grams per second) until the participant indicates verbally that the pain threshold has been reached.
Time Frame: Baseline
Population: One person was erroneously randomized to placebo before they were eligible for randomization and dropped out prior to induction, so they are not considered in this analysis.
Measure: Mean (Full Range); unit: grams per second
Groups:
- Gabapentin + Buprenorphine Taper: Group randomized to Gabapentin + buprenorphine taper in Phase II
- Placebo + Buprenorphine Taper: Group Randomized to Placebo and Buprenorphine Taper in Phase II
Arm/Group | Gabapentin + Buprenorphine Taper | Placebo + Buprenorphine Taper
Number analyzed (Participants) | 13 | 13
grams per second | 284.2 [113.7 to 482.7] | 289.1 [163.6 to 627.3]

6. Secondary Outcome: Mean Score of Current Opioid Measure (COMM)
Description: COMM is a 17 item questionnaire that is used to examine concurrent misuse. The score range is from 0-28. A lower score represents participant showing less aberrant behaviors associates with misuse of option medications, and a higher score represents more aberrant behaviors associated with opioid medical misuse.
Time Frame: Baseline
Population: One person erroneously randomized to placebo before eligible for induction and who never completed buprenorphine induction not considered in this analysis.
Measure: Mean (Full Range); unit: units on a scale
Groups:
- Gabapentin + Buprenorphine Taper: Those randomized to Gabapentin during buprenorphine taper in Phase II after buprenorphine induction.
- Placebo + Buprenorphine Taper: Those randomized to Placebo during buprenorphine taper in Phase II after buprenorphine induction.
Arm/Group | Gabapentin + Buprenorphine Taper | Placebo + Buprenorphine Taper
Number analyzed (Participants) | 13 | 13
units on a scale | 16 [1 to 41] | 15 [5 to 49]

7. Secondary Outcome: Mean Score of PROMIS Physical Function Short Form (PROMIS SF 10) - RAW SCORE PH
Description: The Mean score of Physical Function on PROMIS short form. The global physical health score is a sum of responses to 4 questions. The range is from 4-20. A lower score represents lower physical function.
  The following questions will be asked: In general, how would you rate your physical health? (range is 1-5; 1 represents poor rating in health, 5 represents excellent rating of physical health) To what extent are you able to carry out your everyday physical activities such as walking, climbing stairs, carrying groceries, or moving a chair? (range is 1-5; 1 represents score of not at all, 5 represents score of completely) How would you rate your fatigue on average? (range is 1-5; 1 represents very severe fatigue, and 5 represents no fatigue) How would you rate your pain on average (range is 0-10; 0 represents no pain, 10 represents worst pain imaginable). The pain score is then recoded: 0, no pain = 5; 1, 2, or 3 = 4; 4, 5, or 6 =3; 7, 8, 9 =2;10 =1
Time Frame: baseline
Population: This form was introduced after the first 2 participants had been randomized, so we only have this data for the 24 who were randomized after buprenorphine induction (vs n=26 for other outcome measures). One person was erroneously randomized prior to eligibility for randomization and was not included in calculations for these secondary outcomes.
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Gabapentin + Buprenorphine Taper | Placebo + Buprenorphine Taper
Number analyzed (Participants) | 12 | 12
units on a scale | 10.3 [8 to 14] | 11 [7 to 14]

8. Secondary Outcome: Mean Score Pittsburgh Sleep Quality Index
Description: The PSQI is a 19 item self-report questionnaire that assesses sleep quality over a 1-month time interval. The measure consists of 19 individual items, creating 7 components (time gone to bed, how long it takes to go to sleep, wake up time, hours slept, issues sleeping, total hours slept etc.) that produce one global score. Each item is weighted on a 0-3 interval scale. The global score is calculated by totaling the seven component scores, providing an overall score ranging from 0 to 21, A lower scale is indicative of better sleep quality and higher score represents poor sleep quality.
Time Frame: baseline
Population: One person erroneously randomized not included
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Gabapentin + Buprenorphine Taper | Placebo + Buprenorphine Taper
Number analyzed (Participants) | 13 | 13
units on a scale | 12.5 [4 to 19] | 10.6 [4 to 16]

9. Secondary Outcome: Mean Score of Subjective Opioid Withdrawal Scale (SOWS)
Description: The Subjective Opiate Withdrawal Scale (SOWS) consist of 16 symptoms rated in intensity by patients on a 5-point scale of intensity as follows: 0=not at all, 1=a little, 2=moderately, 3=quite a bit, 4=extremely. The total score is a sum of item ratings, and ranges from 0 to 64.
Time Frame: baseline
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Gabapentin + Buprenorphine Taper | Placebo + Buprenorphine Taper
Number analyzed (Participants) | 13 | 13
units on a scale | 17.3 [0 to 58] | 11.9 [0 to 49]

10. Secondary Outcome: Number of Participants Who Achieved Opioid Cessation Post-taper - 3 Months
Description: Opioid cessation is evidenced as a score of 3 points when summing the following measures: self-report of no opioid use = 1 point; prescription drug monitoring data showing no opioid prescriptions filled in past 30 days = 1 point; and confirmatory negative urine toxicology for a full panel of opioids = 1 point.
Time Frame: Post-taper - 3 months
Population: One person in the Gabapentin + Buprenorphine Taper Arm completed the study buprenorphine taper and were eligible for analysis. Zero persons in the Placebo + Buprenorphine Taper Arm completed the study buprenoprhine taper and were eligible for analysis.
Measure: Count of Participants; unit: Participants
Groups:
- Gabapentin + Buprenorphine Taper - Opioid Cessation 3 Months Post-taper: One person in the Gabapentin + Buprenorphine Taper Arm completed the study buprenorphine taper
- Placebo + Buprenorphine Taper - Opioid Cessation 3 Months Post-taper: Zero persons in the Placebo + Buprenorphine Taper Arm completed the study buprenorphine taper.
Arm/Group | Gabapentin + Buprenorphine Taper - Opioid Cessation 3 Months Post-taper | Placebo + Buprenorphine Taper - Opioid Cessation 3 Months Post-taper
Number analyzed (Participants) | 1 | 0
Participants | 1 | 0

11. Secondary Outcome: Number of Participants Who Achieved Opioid Cessation Post-taper - 6 Months
Description: as for outcome 10
Time Frame: Post-taper - 6 months
Population: One person in the Gabapentin + Buprenorphine Taper Arm completed the study buprenorphine taper, and zero persons in the Placebo + Buprenorphine Taper Arm completed the study buprenorphine taper.
Measure: Count of Participants; unit: Participants
Groups:
- Gabapentin + Buprenorphine Taper - Opioid Cessation 6 Months Post-taper: One person in the Gabapentin + Buprenorphine Taper Arm completed the study buprenorphine taper.
- Placebo + Buprenorphine Taper - Opioid Cessation 6 Months Post-taper: Zero persons in the Placebo + Buprenorphine Taper Arm completed the study buprenorphine taper.
Arm/Group | Gabapentin + Buprenorphine Taper - Opioid Cessation 6 Months Post-taper | Placebo + Buprenorphine Taper - Opioid Cessation 6 Months Post-taper
Number analyzed (Participants) | 1 | 0
Participants | 1 | 0

12. Secondary Outcome: Number of Participants Who Achieved Opioid Cessation Post-taper - 12 Months
Description: as for outcome 10
Time Frame: Post-taper - 12 months
Population: One person in the Gabapentin + Buprenorphine Taper Arm and Zero people in the Placebo + Buprenorphine Taper Arm completed the study buprenorphine taper.
Measure: Count of Participants; unit: Participants
Groups:
- Gabapentin + Buprenorphine Taper - Opioid Cessation 12 Months Post-taper: One person in the Gabapentin + Buprenorphine Taper Arm completed the study buprenorphine taper.
- Placebo + Buprenorphine Taper - Opioid Cessation 12 Months Post-taper: Zero persons in the Placebo + Buprenorphine Taper Arm completed the study buprenorphine taper.
Arm/Group | Gabapentin + Buprenorphine Taper - Opioid Cessation 12 Months Post-taper | Placebo + Buprenorphine Taper - Opioid Cessation 12 Months Post-taper
Number analyzed (Participants) | 1 | 0
Participants | 1 | 0

13. Secondary Outcome: Pain Laboratory Measures - Descending Noxious Inhibitory Control (DNIC) - Average, Baseline
Description: DNIC will be measured as the percent change in PPTh during the cold pressor tasks relative to baseline. A percent increase represents normal functioning of pain inhibitory processes.
Time Frame: Baseline
Population: One person was erroneously randomized to placebo before eligible for randomization, and never completed buprenorphine induction, so they are not considered in this analysis.
Measure: Mean (Full Range); unit: percentage of change
Arm/Group | Gabapentin + Buprenorphine Taper | Placebo + Buprenorphine Taper
Number analyzed (Participants) | 13 | 13
percentage of change | 312.5 [139.5 to 538.7] | 326.4 [178.8 to 631.3]

ADVERSE EVENTS:
Time Frame: 12 months
Groups:
- Phase I - Buprenorphine Initiation: In Phase I, we will determine buprenorphine tolerability using a one-day outpatient buprenorphine initiation protocol up to 16mg sublingually over an 8 hour induction window.
- Phase II - Gabapentin + Buprenorphine: Subjects who tolerate sublingual buprenorphine initiation in Phase I will proceed to Phase II, which will involve randomization to oral gabapentin or placebo, 2 week stabilization period, and up to 8 week buprenorphine tapering period. Those randomized to gabapentin will receive up to 1600mg gabapentin (double blinded) divided three times daily, titrated over the 2 week stabilization period and continued during the buprenorphine tapering period. During the 2 week stabilization period, buprenorphine will also be titrated up to 24mg as needed/tolerated.
- Phase II - Gabapentin + Placebo: Subjects who tolerate sublingual buprenorphine initiation in Phase I will proceed to Phase II, which will involve randomization to oral gabapentin or placebo, 2 week stabilization period, and up to 8 week buprenorphine tapering period. Those randomized to placebo will receive up to 1600mg placebo (double blinded) divided three times daily, titrated over the 2 week stabilization period and continued during the buprenorphine tapering period. During the 2 week stabilization period, buprenorphine will also be titrated up to 24mg as needed/tolerated.
Arm/Group | Phase I - Buprenorphine Initiation | Phase II - Gabapentin + Buprenorphine | Phase II - Gabapentin + Placebo | Phase II - Buprenorphine Taper
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/13 | 0/14 | 0/27
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/13 | 0/14 | 0/27
Other Adverse Events (participants affected / at risk) | 2/27 | 12/13 | 12/14 | 0/27
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I - Buprenorphine Initiation (N=27) | Phase II - Gabapentin + Buprenorphine (N=13) | Phase II - Gabapentin + Placebo (N=14) | Phase II - Buprenorphine Taper (N=27)
Increased Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (7) | 5 (9) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 4 (8) | 4 (7) | 0 (0)
Dry Mouth (General disorders) | 0 (0) | 3 (5) | 4 (6) | 0 (0)
Lower extremity swelling (Blood and lymphatic system disorders) | 0 (0) | 2 (4) | 6 (7) | 0 (0)
Insomnia (General disorders) | 0 (0) | 3 (5) | 4 (8) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 4 (7) | 2 (4) | 0 (0)
Muscle twitching/spasm (Nervous system disorders) | 0 (0) | 3 (3) | 3 (3) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (2) | 3 (5) | 0 (0)
Sedation/sleepiness (General disorders) | 2 (2) | 4 (6) | 2 (4) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-25): https://cdn.clinicaltrials.gov/large-docs/26/NCT02737826/Prot_SAP_000.pdf